CLINICAL TRIAL: NCT04706039
Title: Rapid Diagnosis of COVID-19 by Chemical Analysis of Exhaled Air
Acronym: COVIDAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL20_1148
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2021-07

CONDITIONS: Covid19
Keywords: covid19 diagnostic; Proton Transfer Mass Spectrometer; exhaled air; rapid and non-invasive diagnosis
MeSH Terms: conditions — COVID-19; Fasting | interventions — Sensitivity and Specificity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Outpatients without hospitalisation criteria (Experimental): Symptomatic and asymptomatic outpatient without hospitalisation criteria presenting in a COVID-19 screening centre of the Hospices Civils de Lyon
  Interventions: Diagnostic Test: Performance evaluation (sensitivity and specificity) for COVID-19 diagnosis of the Vocus PTR-TOF process

INTERVENTIONS:
Diagnostic Test: Performance evaluation (sensitivity and specificity) for COVID-19 diagnosis of the Vocus PTR-TOF process — Each patient will be sampled to do a systematic respiratory virus infection screening (SARS-CoV-2 and Flu and RSV). Then each patient will be tested using the Vocus PTR-TOF process.
  A self-answering questionnaire will be used to collect symptomatology information and date of onset of symptoms.

SUMMARY:
Since the start of 2020, the new SARS-CoV-2 coronavirus is causing a real global health crisis.

In France, nasopharyngeal swabs are used to obtain the sample needed for respiratory infection screening. There are three major difficulties with this type of sampling:

I) It is really unpleasant for the patient because the device has to be pushed into the nostril to reach the nasopharynx. It causes some patients to bleed or even feel uncomfortable.

II) It is not easily accepted by children. III) It is dependent on the availability of swabs. Faced with these difficulties linked to the initial sampling, new methods are being studied to enable a rapid and non-invasive diagnosis of COVID-19 based on the instantaneous identification of metabolites or volatile organic compounds (VOCs).

Due to their sensitivity and the wealth of information that can be provided, the most promising techniques are based on mass spectrometry coupled with a soft ionisation system. For example, on-line exhaled air analysis is capable of detecting a very large number of VOCs. Various tests on metabolites in the exhaled air have already been carried out without being totally conclusive because the existing instruments suffer from various limitations:

I) poor repeatability/accuracy in the chemical characterisation of exhaled air ; II) too high specificity (detection of only part of the emitted compounds); III) too limited sensitivity; IV) and poor adaptation to be deployed in a clinic.

In order to overcome these various limitations, we propose the use of a new generation of mass spectrometer: Vocus PTR-TOF. The Vocus PTR-TOF is a Proton Transfer Mass Spectrometer (PTR-MS) developed for the detection, in real time, of trace VOCs in industrial environments, laboratories or directly in the environment. This new generation of instrument offers the following advantages:

I) unequalled sensitivity :

II) a robust ionisation system not affected by environmental conditions (relative humidity...) ; III) a high mass resolution allowing precise identification of compounds ; IV) a compact and durable architecture allowing deployment in a constrained environment such as hospital, airport… The sensitivity and speed of measurement allow the expiration process to be monitored in real time, bringing an additional dimension to the measurement and the chances of success.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic and asymptomatic outpatient without hospitalisation criteria
* No medical contraindications to nasopharyngeal swabbing (deviation of the nasal septum, epistaxis, anticoagulant treatment).
* Patient able to blow into the test device
* Patients or parents with parental authority who have been informed of the study and have not objected to participating in it

Exclusion Criteria:

* Major subject under guardianship or curatorship or unable to consent to study.
* Subject under safeguard of justice
* Minor patient (age < 6 years).

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4600 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the COVID-19 diagnostic using the Vocus PTR-TOF process. | At the inclusion visit
  Study of the sensitivity of the exhaled air test in comparison to the reference diagnostic RT-PCR on nasopharyngeal swab. We will use the results of the RT-PCR as reference to compare the results of the Vocus PTR-TOF process.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de prélèvement COVID-19 HCL et Métropole de Lyon, Lyon, France